CLINICAL TRIAL: NCT07004491
Title: Comparison Of Different Physiotherapy Methods In People With Non-Specific Neck Pain
Acronym: Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3746
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Neck Pain
Keywords: Non specific neck pain; physiotherapy applicaitons; pain
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First Intervention (Experimental): 5 minutes of Ultrasound, 20 minutes of Transcutaneous Electrical Nerve Stimulation (TENS) and hot pack application will be applied.
  Interventions: Other: Conventional therapy
- Second Intervention (Experimental): In addition to 5 minutes of Ultrasound, 20 minutes of Transcutaneous Electrical Nerve Stimulation (TENS) and hot pack application, Mulligan mobilization technique will be applied. Continuous apophyseal shifting technique will be applied as mobilization. Mobilization will be applied in 3 sets of 4-5 repetitions.
  Interventions: Other: Conventional therapy+ Mulligan mobilization
- Third Intervention (Experimental): In addition to 5 minutes of Ultrasound, 20 minutes of Transcutaneous Electrical Nerve Stimulation (TENS) and hot pack application, Graston treatment will be applied to the upper and lower trapezius, rhomboid major and minor muscles for 5 minutes.
  Interventions: Other: Conventional therapy+ Graston

INTERVENTIONS:
Other: Conventional therapy — Ultrasound, Transcutaneous Electrical Nerve Stimulation (TENS) and hot pack application
  Arms: First Intervention
Other: Conventional therapy+ Mulligan mobilization — Conventional therapy+ Mulligan mobilization
  Arms: Second Intervention
Other: Conventional therapy+ Graston — Conventional therapy+ Graston application
  Arms: Third Intervention

SUMMARY:
The study will include 45 people between the ages of 25-55 with non-specific neck pain. The patients will be randomly divided into three groups. Group 1 will receive 5 minutes of ultrasound, 20 minutes of transcutaneous electrical nerve stimulation (TENS), and hot pack application. Group 2 will receive 5 minutes of ultrasound, 20 minutes of transcutaneous electrical nerve stimulation (TENS), and hot pack application in addition to the Mulligan mobilization technique. Group 3 will receive 5 minutes of ultrasound, 20 minutes of transcutaneous electrical nerve stimulation (TENS), and hot pack application in addition to graston treatment for 5 minutes to the upper and lower trapezius, rhomboid major and minor muscles.

DETAILED DESCRIPTION:
The study will include 45 people between the ages of 25-55 with non-specific neck pain. The patients will be randomly divided into three groups. Group 1 will receive 5 minutes of ultrasound, 20 minutes of transcutaneous electrical nerve stimulation (TENS), and hot pack application. Group 2 will receive 5 minutes of ultrasound, 20 minutes of transcutaneous electrical nerve stimulation (TENS), and hot pack application in addition to the Mulligan mobilization technique. Group 3 will receive 5 minutes of ultrasound, 20 minutes of transcutaneous electrical nerve stimulation (TENS), and hot pack application in addition to graston treatment for 5 minutes to the upper and lower trapezius, rhomboid major and minor muscles. The patients will receive treatments 3-4 times a week for 4 weeks, for a total of 10 sessions. VAS, neck joint range of motion, functional status and disability level neck pain and disability scale and SF-36 will be used as evaluation measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with non-specific neck pain by a doctor
* aged between 25-55
* who have had pain in their neck for at least 2 weeks will be included in the study.

Exclusion Criteria:

* Neurological disease
* Manual therapy contraindication such as osteoporosis, spinal infection
* Spondyloarthropathy, disc herniation
* People with contraindications to the Graston technique such as neoplastic disorders, anticoagulant drug use, uncontrolled hypertension or general infection will not be included in the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-07-26 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Visucal Analog scale | 10 minutes
  The Visual Analog Scale (VAS) (0-10 cm), which is found to be valid, reliable and sensitive in patients with neck pain, will be used to assess pain. O means no pain; 10 means severe pain.
Joint range of motion | 20 minutes
  The patients' neck joint range of motion will be measured with a standard goniometer.
Quality of life (SF-36) | 15 minutes
  SF-36 will be used to assess the participants' quality of life. The 36-question questionnaire is divided into 8 groups: physical role functioning, emotional role functioning, bodily pain, energy, social role functioning, mental health and general health perception. Each category is scored between 0-100 and higher scores indicate better quality of life
The neck disability scale | 15 minutes
  Functional status and disability level will be assessed with the neck pain and disability scale.The neck disability scale will be used to assess how the participants' daily lives are affected by neck pain. The total score of the scale ranges from 0 to 35, with higher scores indicating higher levels of disability

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, Assoc. Prof., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We can share IPD if it is need.

REFERENCES:
- [Result] Mahmood T, Afzal W, Ahmad U, Arif MA, Ahmad A. Comparative effectiveness of routine physical therapy with and without instrument assisted soft tissue mobilization in patients with neck pain due to upper crossed syndrome. J Pak Med Assoc. 2021 Oct;71(10):2304-2308. doi: 10.47391/JPMA.03-415. PMID 34974559
- See also: Comparative effectiveness of routine physical therapy with and without instrument assisted soft tissue mobilization in patients with neck pain due to upper crossed syndrome. — https://pubmed.ncbi.nlm.nih.gov/34974559/